CLINICAL TRIAL: NCT03444298
Title: A Phase II Randomized, Double Blinded, Placebo-controlled Study of Gamma Tocopherol-enriched Supplement on Lower Airway Responses to Inhaled Wood Smoke in Healthy Adults
Brief Title: A Study of Gamma Tocopherol-enriched Supplement on Lower Airway Responses to Inhaled Wood Smoke in Healthy Adults
Acronym: SmokeyT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-2303; 5R01ES025124 (NIH)
Record Dates: First submitted 2018-01-31; First posted 2018-02-23 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Airway Inflammation; Asthma
MeSH Terms: conditions — Asthma | interventions — gamma-Tocopherol; Vitamin E

STUDY DESIGN:
Intervention Model Description: Subjects will be allocated to begin the first period of the crossover study with placebo or gamma tocopherol treatment using permuted block randomization with a block size of 4 (2 placebo, 2 gamma tocopherol for the first treatment period of the protocol).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization schedule will be generated by the biostatistician and provided to the investigational pharmacy. Only the biostatistician and the pharmacist will have access to the randomization schedule.
  Participants will consume 1400 mg of γT-enriched supplement or matching placebo once daily for 7 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo first, then Gamma Tocopherol (Placebo Comparator): Participants that are randomized to placebo treatment will take a short treatment course of Neutral Oil followed by chamber exposure with wood smoke particulate. After a 4-week washout period, participants will cross over to the gamma Tocopherol (active) treatment group.
  Interventions: Drug: Gamma Tocopherol; Drug: Placebo
- GammaTocopherol first, then Placebo (Active Comparator): Participants that are randomized γT treatment will take a short treatment course of gamma Tocopherol followed by chamber exposure with WSP. After a 4-week washout period, participants will cross over to the placebo treatment group.
  Interventions: Drug: Gamma Tocopherol; Drug: Placebo

INTERVENTIONS:
Drug: Gamma Tocopherol — Each dose consists of two (700 mg) capsules by mouth once daily for a total of 7 days.
  Other Names: Vitamin E
Drug: Placebo — Each dose consists of two capsules by mouth once daily for a total of 7 days.
  Other Names: Neutral oil

SUMMARY:
Purpose: To determine the efficacy of 1400 mg gamma tocopherol-enriched supplement for mitigating inhaled wood smoke particle-induced airway inflammation in healthy adults with no more than mild asthma.

DETAILED DESCRIPTION:
Particulate matter (PM) is a leading cause of respiratory tract and cardiovascular disease in the United States and world-wide. Wood smoke particles (WSP) derived from wildland and other fires account for a significant fraction of ambient air PM. Health effects associated with WSP include acute bronchitis, asthma exacerbation, pneumonia, cough and systemic inflammation. While these effects are seen in both healthy and asthmatic individuals, many studies indicate that asthmatics have increased susceptibility to the effects of WSP. The investigators have developed a 500 μg/m3 WSP exposure protocol (levels similar to those encountered by firefighters and residents in close proximity to wildland burn sites) that induces airway and systemic inflammation in healthy volunteers. As with other pollutants, these inflammatory responses modulate non-specific bronchial reactivity (NSBR), inflammatory cell recruitment to the airways (primarily neutrophils), and potentially cardiovascular function.

The investigators have focused on gamma tocopherol (γT) as a nutritional intervention to prevent inflammatory responses to air pollutants such as WSP. Building on animal and in vitro preclinical studies, the investigators have established that 1400 mg/day of oral γT-enriched supplement for 7 and 14 days in healthy volunteers and mild asthmatics, respectively, inhibited neutrophil influx into the airways, reduced production of sputum mucins, and improved mucociliary clearance following challenge with inhaled endotoxin, another common component of PM. The findings occurred in the context of significantly increased plasma concentrations of γT and its active metabolite 2,7,8-trimethyl-2-(β-Carboxy-Ethyl)-6-Hydroxychroman (γ-CEHC). Given the findings in these early phase clinical trials, γT supplementation is an attractive approach to prevent WSP-induced adverse health effects. The investigators propose to use γT supplementation in a human model of WSP inhalation to mitigate key features of airway inflammation: inflammatory cell recruitment, production of inflammatory cytokines and mucous, and changes in airway physiology.

Gamma tocopherol will be administered in softgel form, with each softgel containing 700 mg of tocopherols, 89.5% of which is d-gamma tocopherol. Subjects will consume two softgels by mouth once daily for 7 days. This dosing regimen was chosen based on the results of the investigators' previous early phase clinical trials examining the impact of gamma tocopherol on lipopolysaccharide (LPS) -induced airway inflammation in healthy adults and adults with asthma. These studies tested a 7 and 14 day course of treatment, respectively, and found similar plasma concentrations of γT and active metabolites in both studies. Furthermore, the investigators showed in both studies that γT significantly reduced LPS-induced sputum neutrophilia compared to placebo. Based on the previous findings, the investigators will now study the efficacy of γT for mitigating WSP-induced airway inflammation.

January 2022 update: The existing, custom source of gamma tocopherol expired during the protocol paused period during Covid. The Gamma t is replaced by Gamma E Gems, manufactured by Carlson Labs, each capsule with 577mg of gamma tocopherol, based on Certificate of Analysis. Subjects will continue to ingest 2 capsules at each dosing, for a total dose of 1154mg. The safflower oil placebo is replaced with a neutral oil capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years, inclusive, of both genders
2. Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy
3. Forced expiratory volume at one second (FEV1) of at least 75% of predicted (without use of bronchodilating medications for 12 hours), consistent with lung function of persons with no more than mild intermittent or mild persistent asthma.
4. Oxygen saturation of <93% and blood pressure within the following limits: (Systolic between 150-85 mmHg, Diastolic between 90-50 mmHg).
5. Ability to provide an induced sputum sample.
6. Subject must demonstrate a ≥10% increase in sputum neutrophils following inhaled WSP exposure, when compared to baseline sputum (to be completed in a separate protocol).
7. Ability/willingness to discontinue inhaled corticosteroids, montelukast, and cromolyn for 2 weeks without increased symptoms or increased need for beta agonist rescue medication prior to screening and through the course of the study.

Exclusion Criteria

Patients who meet any of these criteria are not eligible for enrollment as study participants:

1. Clinical contraindications:

   1. Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections/immunodeficiency.
   2. Viral upper respiratory tract infection within 4 weeks of challenge.
   3. Any acute infection requiring antibiotics within 4 weeks of exposure or fever of unknown origin within 4 weeks of challenge.
   4. Abnormal physical findings at the baseline visit, including but not limited to abnormalities on auscultation, temperature of 37.8° C, Systolic BP > 150mm Hg or < 85 mm Hg; or Diastolic BP > 90 mm Hg or < 50 mm Hg, or pulse oximetry saturation reading less than 93%.
   5. Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
   6. Moderate or severe asthma
   7. Exacerbation of asthma more than 2x/weeks which would be characteristic of a person with moderate or severe persistent asthma as outlined in the current National Asthma Education and Prevention Program (NAEPP) guidelines for diagnosis and management of asthma
   8. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person with moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma (not to include prophylactic use of albuterol prior to exercise).
   9. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for the diagnosis and management of asthma.
   10. History of intubation for asthma
   11. If there is a history of allergic rhinitis, subjects must be asymptomatic of allergic rhinitis at the time of study enrollment.
   12. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
   13. Cigarette smoking > 1 pack per month
   14. Unwillingness to use reliable contraception if sexually active (IUD, birth control pills/patch, condoms).
   15. Abnormal prothrombin time (PT) or activated partial thromboplastin time (aPTT) values at screening or during the treatment period. Normal values will be those published by the clinical lab (Labcorp, INC).
   16. Use of immunosuppressive or anticoagulant medications including routine use of NSAIDS. Oral contraceptives are acceptable, as are Antidepressants and other medications may be permitted if, in the opinion of the investigator, the medication will not interfere with the study procedures or compromise safety and if the dosage has been stable for 1 month.
   17. Orthopedic injuries or impediments that would preclude bicycle or treadmill exercise.
   18. Inability to avoid NSAIDS, Multivitamins, Vitamin C or E or herbal supplements.
   19. Allergy/sensitivity to study drugs or their formulations
   20. Known hypersensitivity to methacholine or to other parasympathomimetic agents
   21. Unwillingness to avoid coffee, tea, cola drinks, chocolate, or other foods containing caffeine after midnight on the days that methacholine challenge testing is to be performed.
2. Pregnant/nursing women and children (< 18 years as this is age of majority in North Carolina) will also be excluded since the risks associated with woodsmoke exposure to the fetus or child, respectively, are unknown and cannot be justified for this non-therapeutic protocol. Individuals over 45 years of age will not be included due to the increased possibility of co-morbidities and need for prohibited medications.
3. Inability or unwillingness of a participant to give written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Peden, MD, Principal Investigator — UNC
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burbank AJ, Duran CG, Almond M, Wells H, Jenkins S, Jiang Q, Yang C, Wang T, Zhou H, Hernandez ML, Peden DB. A short course of gamma-tocopherol mitigates LPS-induced inflammatory responses in humans ex vivo. J Allergy Clin Immunol. 2017 Oct;140(4):1179-1181.e4. doi: 10.1016/j.jaci.2017.04.030. Epub 2017 May 12. No abstract available. PMID 28506847
- [Background] Hernandez ML, Wagner JG, Kala A, Mills K, Wells HB, Alexis NE, Lay JC, Jiang Q, Zhang H, Zhou H, Peden DB. Vitamin E, gamma-tocopherol, reduces airway neutrophil recruitment after inhaled endotoxin challenge in rats and in healthy volunteers. Free Radic Biol Med. 2013 Jul;60:56-62. doi: 10.1016/j.freeradbiomed.2013.02.001. Epub 2013 Feb 9. PMID 23402870
- [Background] Wiser J, Alexis NE, Jiang Q, Wu W, Robinette C, Roubey R, Peden DB. In vivo gamma-tocopherol supplementation decreases systemic oxidative stress and cytokine responses of human monocytes in normal and asthmatic subjects. Free Radic Biol Med. 2008 Jul 1;45(1):40-9. doi: 10.1016/j.freeradbiomed.2008.03.002. Epub 2008 Mar 12. PMID 18405673
- [Background] Burbank AJ, Duran CG, Pan Y, Burns P, Jones S, Jiang Q, Yang C, Jenkins S, Wells H, Alexis N, Kesimer M, Bennett WD, Zhou H, Peden DB, Hernandez ML. Gamma tocopherol-enriched supplement reduces sputum eosinophilia and endotoxin-induced sputum neutrophilia in volunteers with asthma. J Allergy Clin Immunol. 2018 Apr;141(4):1231-1238.e1. doi: 10.1016/j.jaci.2017.06.029. Epub 2017 Jul 20. PMID 28736267
- [Result] Peden DB, Almond M, Brooks C, Robinette C, Wells H, Burbank A, Hernandez M, Hinderliter A, Caughey M, Jiang Q, Wang Q, Li H, Zhou H, Alexis N. A pilot randomized clinical trial of gamma-tocopherol supplementation on wood smoke-induced neutrophilic and eosinophilic airway inflammation. J Allergy Clin Immunol Glob. 2023 Oct 5;2(4):100177. doi: 10.1016/j.jacig.2023.100177. eCollection 2023 Nov. PMID 37876758

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven persons completed the study. The original gT dose was 1 dose every 12 hours x 4 (n=4 volunteers), but was ineffective in another study, so dosing was increased to 7 daily doses (n=4 volunteers). The gT expired during an 18 month pause for COVID-19 and could not be replaced, and a similarly potent commercially available gT-enriched preparation for 7 daily doses was then used for the final 3 persons. An intent-to-treat analysis of primary end points for all completed volunteers was used.
Groups:
- Placebo First, Then Gamma Tocopherol: Participants that are randomized to placebo treatment will take a short treatment course of Neutral Oil followed by chamber exposure with wood smoke particulate. After a 4-week washout period, participants will cross over to the gamma Tocopherol (active) treatment group.
  Gamma Tocopherol (gT): Each dose consists of two (700 mg) capsules by mouth once daily for a total of 7 days.
  Placebo: Each dose consists of two capsules by mouth once daily for a total of 7 days.
Period: Period 1 (Dosing Followed by Exposure)
Arm/Group | Placebo First, Then Gamma Tocopherol | GammaTocopherol First, Then Placebo
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0
Period: Washout (>/= 4 Weeks)
Arm/Group | Placebo First, Then Gamma Tocopherol | GammaTocopherol First, Then Placebo
Started | 7 | 9
Completed | 4 | 7
Not Completed | 3 | 2
Period: Period 2 (Dosing Followed by Exposure)
Arm/Group | Placebo First, Then Gamma Tocopherol | GammaTocopherol First, Then Placebo
Started | 4 | 7
Completed | 4 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Gamma Tocopherol | GammaTocopherol First, Then Placebo | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 00 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 3 | 8 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Sputum % Polymorphonuclear Neutrophils (PMN) With Wood Smoke Particulate (WSP) Exposure
Description: A comparison of the WSP-induced change in sputum % PMNs (Post-WSP sputum - Pre-WSP sputum) during gamma tocopherol treatment with the WSP-induced change in sputum % PMNs during placebo treatment.
Time Frame: baseline, and 4 hours post exposure
Population: Data are reported for participants who completed both arms and provided adequate sputum samples.
Measure: Mean (Standard Deviation); unit: percent PMNs
Groups:
- GammaTocopherol: Participants receive two (700 mg) capsules by mouth once daily for a total of 7 days.
- Placebo: Participants receive two placebo capsules by mouth once daily for a total of 7 days.
Arm/Group | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11
percent PMNs | 18.00 (20.89) | 14.75 (17.98)
Statistical Analysis 1: Comparison: GammaTocopherol vs Placebo; Test type: Superiority; p = 0.67, t-test, 2 sided — The a priori threshold for statistical significance is <0.05

2. Primary Outcome: Change in Sputum % PMNs With WSP Exposure
Description: as for outcome 1
Time Frame: baseline, and 24 hours post exposure
Population: Data are reported for participants who completed both arms and provided adequate sputum samples as outlined for each arm. Three participants did not have adequate sputum at 24 hours after active treatment.
Measure: Mean (Standard Deviation); unit: percent PMNs
Arm/Group | GammaTocopherol | Placebo
Number analyzed (Participants) | 8 | 11
percent PMNs | 39.87 (20.59) | 29.35 (28.30)
Statistical Analysis 1: Comparison: GammaTocopherol vs Placebo; Test type: Superiority; p = 0.43, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05

3. Secondary Outcome: Change in Absolute PMN Count (ANC) in Sputum With WSP Exposure
Description: A comparison of the WSP-induced change in sputum ANC (Post-WSP sputum - Pre-WSP sputum) during gamma tocopherol treatment with the WSP-induced change in sputum ANC during placebo treatment.
Time Frame: baseline, and 4 hours post exposure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: PMNs per mg sputum
Arm/Group | GammaTocopherol | Placebo
Number analyzed (Participants) | 8 | 11
PMNs per mg sputum | 8.58 (150.6) | -20.51 (160.6)
Statistical Analysis 1: Comparison: GammaTocopherol vs Placebo; Test type: Superiority; p = 0.27, t-test, 2 sided — The a priori threshold for statistical significance is <0.05

4. Secondary Outcome: Change in Absolute PMN Count (ANC) in Sputum With WSP Exposure
Description: as for outcome 3
Time Frame: baseline, and 24 hours post exposure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: PMNs per mg sputum
Arm/Group | GammaTocopherol | Placebo
Number analyzed (Participants) | 8 | 11
PMNs per mg sputum | 104.7 (146.5) | 96.7 (156.2)
Statistical Analysis 1: Comparison: GammaTocopherol vs Placebo; Test type: Superiority; p = 0.92, t-test, 2 sided — The a priori threshold for statistical significance is <0.05

5. Post Hoc Outcome: Percent Eosinophils in Sputum
Description: A comparison of the WSP-induced sputum % eosinophils versus predosing values with gamma tocopherol and placebo treatment.
Time Frame: up to 24 hours
Population: Data are reported for participants who completed both arms and provided adequate sputum samples.
Measure: Mean (Standard Deviation); unit: percent eosinophils
Groups:
- Pre-Dosing: Pre-dose, pre-challenge baseline data
Arm/Group | Pre-Dosing | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11 | 11
percent eosinophils
  4 Hours | 0.07 (0.04) | 0.04 (0.08) | 2.3 (1.6)
  24 Hours: number analyzed (Participants) | 11 | 8 | 11
  24 Hours | 0.07 (0.04) | 0.26 (0.15) | 0.39 (0.33)
Statistical Analysis 1: Comparison: Pre-Dosing vs GammaTocopherol; Test type: Superiority; p = 0.99, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Pre-Dosing vs Placebo; Test type: Superiority; p = 0.04, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05

6. Post Hoc Outcome: Eosinophils Per mg Sputum
Description: A comparison of the WSP-induced sputum eosinophils after gamma tocopherol and placebo pre dosing values.
Time Frame: up to 24 hours
Population: Data are reported for participants who completed both arms and provided adequate sputum samples.
Measure: Mean (Standard Deviation); unit: Cells per mg (eosinophils)
Arm/Group | Pre-Dosing | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11 | 11
Cells per mg (eosinophils)
  4 Hours | 0.17 (0.33) | 0.20 (0.52) | 7.10 (12.33)
  24 Hours: number analyzed (Participants) | 11 | 8 | 11
  24 Hours | 0.17 (0.33) | 1.15 (2.11) | 1.02 (2.70)
Statistical Analysis 1: Comparison: Pre-Dosing vs GammaTocopherol; Test type: Superiority; p = 0.98, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Pre-Dosing vs Placebo; Test type: Superiority; p = 0.02, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05

7. Post Hoc Outcome: Interleukin-1 Beta (IL-1β) in Sputum
Description: The IL-1β concentration will be determined in each sputum sample by immunoassay
Time Frame: up to 24 hours
Population: Data are reported for participants who completed both arms and provided adequate sputum samples.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pre-Dosing | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11 | 11
pg/mL
  4 Hours | 798.3 (497.1) | 674.2 (494.9) | 654.4 (438.3)
  24 Hours | 798.3 (497.1) | 469.6 (237.4) | 675.2 (630.6)
Statistical Analysis 1: Comparison: Pre-Dosing vs GammaTocopherol vs Placebo; Test type: Superiority; p = 0.84, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05

8. Post Hoc Outcome: Interleukin-6 (IL-6) in Sputum
Description: The IL-6 concentration will be determined in each sputum sample by immunoassay
Time Frame: up to 24 hours
Population: Data are reported for participants who completed both arms and provided adequate sputum samples.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pre-Dosing | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11 | 11
pg/mL
  4 Hours | 458.0 (492.3) | 384.8 (440.2) | 277.5 (255.5)
  24 Hours | 458.0 (492.3) | 207.0 (171.6) | 281.3 (338.0)
Statistical Analysis 1: Comparison: Pre-Dosing vs GammaTocopherol vs Placebo; Test type: Superiority; p = 0.59, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05

9. Post Hoc Outcome: Interleukin-8 (IL-8) in Sputum
Description: The IL-8 concentration will be determined in each sputum sample by immunoassay
Time Frame: up to 24 hours
Population: Data are reported for participants who completed both arms and provided adequate sputum samples.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pre-Dosing | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11 | 11
pg/mL
  4 Hours | 30850 (28306) | 31724 (37505) | 25432 (23198)
  24 Hours | 30850 (28306) | 17180 (13083) | 36739 (60134)
Statistical Analysis 1: Comparison: Pre-Dosing vs GammaTocopherol vs Placebo; Test type: Superiority; p = 0.83, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05

10. Post Hoc Outcome: Tumor Necrosis Factor-alpha (TNF-a)
Description: The TNF-a concentration will be determined in each sputum sample by immunoassay
Time Frame: up to 24 hours
Population: Data are reported for participants who completed both arms and provided adequate sputum samples.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pre-Dosing | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11 | 11
pg/mL
  4 Hours | 35.67 (25.88) | 127.7 (342.7) | 25.18 (20.84)
  24 Hours | 35.67 (25.88) | 13.77 (12.63) | 29.23 (26.18)
Statistical Analysis 1: Comparison: Pre-Dosing vs GammaTocopherol vs Placebo; Test type: Superiority; p = 0.51, Mixed Models Analysis — The a priori threshold for statistical significance is <0.05

11. Post Hoc Outcome: Alpha Tocopherol in Blood
Description: The alpha tocopherol concentration will be determined in blood samples by high-performance liquid chromatography (HPLC).
Time Frame: Baseline immediately before WSP challenge
Population: Data are reported for participants who completed both arms.
Measure: Mean (Standard Deviation); unit: microM
Arm/Group | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11
microM | 22.54 (10.17) | 24.58 (3.40)
Statistical Analysis 1: Comparison: GammaTocopherol vs Placebo; Test type: Superiority; p = 0.48, t-test, 2 sided — The a priori threshold for statistical significance is <0.05

12. Post Hoc Outcome: 2, 7,8-trimethyl-2S-(G-carboxyethyl)-6-hydroxychromane (g-CEHC) in Blood
Description: The 2, 7,8-trimethyl-2S-(g-carboxyethyl)-6-hydroxychromane (g-CEHC) concentration will be determined in blood samples by high-performance liquid chromatography (HPLC).
Time Frame: Baseline immediately before WSP challenge
Population: Data are reported for participants who completed both arms.
Measure: Mean (Standard Deviation); unit: microM
Arm/Group | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11
microM | 1.912 (2.021) | 0.084 (0.08)
Statistical Analysis 1: Comparison: GammaTocopherol vs Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided — The a priori threshold for statistical significance is <0.05

13. Post Hoc Outcome: GammaTocopherol in Blood
Description: The gamma tocopherol concentration will be determined in blood samples by high-performance liquid chromatography (HPLC).
Time Frame: Baseline immediately before WSP challenge
Population: Data are reported for participants who completed both arms.
Measure: Mean (Standard Deviation); unit: microM
Arm/Group | GammaTocopherol | Placebo
Number analyzed (Participants) | 11 | 11
microM | 32.60 (7.45) | 4.64 (1.71)
Statistical Analysis 1: Comparison: GammaTocopherol vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided — The a priori threshold for statistical significance is <0.05

ADVERSE EVENTS:
Time Frame: From the time a participant signed consent through completion of the second intervention, a total of up to 5 months.
Groups:
- GammaTocopherol: Each dose consists of two (700 mg) capsules by mouth once daily for a total of 7 days.
- Placebo: Each dose consists of two placebo capsules by mouth once daily for a total of 7 days.
Arm/Group | GammaTocopherol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 8/13 | 7/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GammaTocopherol (N=13) | Placebo (N=14)
Gastrointestinal Distress (Gastrointestinal disorders) | 7 (8) | 2 (2)
Headache (General disorders) | 2 (2) | 3 (3)
Viral Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash on both inner arms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1) | 0 (0)
Pinched Nerve in Neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nosebleed (Vascular disorders) | 1 (1) | 0 (0)
Unusual Fatigue or Tiredness (General disorders) | 1 (1) | 1 (1)
Premature Ventricular Contraction (Cardiac disorders) | 1 (1) | 0 (0)
Bruise at Venipuncture Site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Menstrual Cramps (General disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Heart Rate Incease Greater than 75 Percent During Exercise (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT03444298/Prot_SAP_000.pdf